CLINICAL TRIAL: NCT03676855
Title: Comparison Between Bladder Dissection Before and After Uterine Incision in Cesarean Section for Morbidly Adherent Placenta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed abd elfatah elsenity, Lecturer of obs and gyn atainshams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWA000017585MD361/2017
Record Dates: First submitted 2018-08-26; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Morbidly Adherent Placenta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bladder dissection before uterine incision (Active Comparator)
  Interventions: Procedure: bladder dissection
- bladder dissection after uterine incision (Experimental)
  Interventions: Procedure: bladder dissection

INTERVENTIONS:
Procedure: bladder dissection — Comparison between bladder dissection at the beginning of cesarean section For morbidly adherent placenta and between delaying dissection until planning for cesarean hysterectomy

SUMMARY:
Comparison between bladder dissection at the beginning of cesarean section For morbidly adherent placenta and between delaying dissection until planning for cesarean hysterectomy

ELIGIBILITY:
Inclusion Criteria:

1. Women with BMI at or under 35 Kg/m2.
2. Women having previous two cesarean section or more.
3. Women with gestational age more than 32 weeks with viable fetus.
4. Women with any degree of placenta previa .
5. Patient with morbidly adherent placenta on cesarean scar only.

Exclusion Criteria:

1. Patient who are haemodynamically unstable before skin incision.
2. Patient with clinically evident intraamniotic infection.
3. Patient with previous history of bladder injury .

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-31 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Operative time | icluding all cs over the period of one year
  of whole cs
Blood loss | icluding all cs over the period of one year
  through counting soaked towels and weighting them before and after being soaked considering the difference in grams as the calculated blood loss and calculating blood in the suction reservoir and comparing pre and post operative Hb level also haemotacrit level and number of units of packed RBCs transfused
- Incidence of urological | during cs and post operative delayed complication icluding all cs over the period of one year
  - Incidence of urological injuries discovered intraoperative and procedure needed to repair or as a late complication as fistula formation.

SECONDARY OUTCOMES:
Neonatal APGAR score | after delivery of the baby during the 1st 15 minutes
  Neonatal APGAR score
Time taken to create bladder flap | from the start of bladder dissection icluding all cs over the period of one year
  from the start of bladder dissection
3 months post operative filling cystometry | 3 months post operative
  3 months post operative filling cystometry

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes